CLINICAL TRIAL: NCT05646628
Title: The Impact of Comorbid Chronic Pain on Older Adults With Depression in Behavioral Activation: A Nested Qualitative Sub-Study of Participants in the BASIL+ Trial
Brief Title: The Impact of Comorbid Chronic Pain on Older Adults With Depression in Behavioral Activation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Teesside University (Other)
Collaborators: University of York (Other)
Responsible Party: Principal Investigator, Alexandra Carne, Principle Investigator, Teesside University
Other Study IDs: 293203; ISRCTN63034289 (Registry Identifier: ISRCTN Registry)
Record Dates: First submitted 2022-11-28; First posted 2022-12-12 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Chronic Pain; Depression
Keywords: Behavioral Activation; Older Adults
MeSH Terms: conditions — Chronic Pain; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Older adults (aged 65 years and over) enrolled in the BASIL+ trial randomized to receive the intervention (collaborative care focusing on behavioral activation) and confirmed as having chronic pain
  Interventions: Behavioral: Qualitative Interviews

INTERVENTIONS:
Behavioral: Qualitative Interviews — Semi-structured Qualitative Interviews

SUMMARY:
This qualitative nested sub-study will aim to explore how chronic pain (as defined as pain lasting for more than 3 months) impacts older adults' depression and treatment in a brief psychological therapy of behavioral activation (BA)

DETAILED DESCRIPTION:
The BASIL + trial (Behavioral Activation in Social Isolation) is a National Institute of Health Research (NIHR) funded and approved trial sponsored by Tees, Esk and Wear Valleys NHS Foundation Trust (TEWV) and led by the University of York in the United Kingdom (UK).

Behavioral Activation (BA) is a type of support that may be beneficial for individuals who suffer from social isolation and/ or depression symptoms. BA assists in the continuation or introduction of activities that are significant to patients. These exercises may be beneficial to both physical and emotional health.

The BASIL+ study aims to find out if BA helps reduce or prevent depression and loneliness in older adults who have ongoing health conditions during isolation in the pandemic due to COVID-19.

Chronic pain affects approximately 50-60% of UK older adults and often coexists with depression. This comorbid indication affects approximately 13% of older adults. The literature on the impact of pain on depression outcomes has been steadily rising. Patients who suffer from depression with comorbid pain report significantly lower benefits, including less relief from depressive symptoms and limits the effectiveness of collaborative care for older adults with depression in the US. The collaborative care focused on antidepressant therapy and problem-solving therapy. Together, these findings suggest that pain may be a potential barrier to depression treatment response. It is unknown, however, how chronic pain impacts depression and the treatment of BA.

This sub-study nested in the BASIL+ trial provides an opportunity to explore how chronic pain impacts depression and the treatment they received

ELIGIBILITY:
Inclusion Criteria:

1. Previously provided optional consent to participate in a qualitative study as part of the BASIL+ trial
2. Not enrolled or offered to take part in any other qualitative study linked with the BASIL+ trial (i.e, the nested BASIL+ qualitative study or the therapeutic alliance sub-study)
3. Suffering chronic pain. This will be assumed by individual scores on the (short-from 12) SF-12 and EuroQoal 5th Edition (EQ-5D) at baseline in the BASIL + trial. Patients who have responded as "moderate, quite a bit or extremely" on question 8 of the SF-12 at baseline and/or responded as having "moderate or extreme pain or discomfort" on the EQ-5D question 4 at baseline will be "assumed" to experiencing some level of pain. A further 2 telephone screening questions by the PI of this sub-study (Alexandra Carne) will assess how often patients have pain and how pain limits their life/work activities in the last 3 months. This will confirm the presence of chronic pain.
4. Participants will have had either a 'favourable' or 'non' favourable' response to treatment. This is defined as having a change of 0.5 SD on the PHQ-9 from baseline to the primary outcome point at 3 months.

Exclusion Criteria:

1. Does not fulfill the inclusion criteria

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Participants will be aged 65 years and older who have depression and were randomized in the BASIL + trial to receive the intervention (collaborative care focusing on behavioral activation) and have been identified as having persistent pain. To ensure maximum diversity, a range of ages, gender, ethnicities and deprivation will be included.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2022-11-28 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Qualitative interview account | July-2022- July2023
  Semi-structured interviews with a topic guide underpinned by a phenomenological framework will be used

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra S Carne, PhD Student, Principal Investigator — Teesside University
Locations (1):
- Teesside University, Middlesbrough, United Kingdom

REFERENCES:
- [Background] Burke L, Littlewood E, Gascoyne S, McMillan D, Chew-Graham CA, Bailey D, Sloan C, Fairhurst C, Baird K, Hewitt C, Henry A, Ryde E, Shearsmith L, Coventry P, Crosland S, Newbronner E, Traviss-Turner G, Woodhouse R, Clegg A, Gentry T, Hill A, Lovell K, Dexter Smith S, Webster J, Ekers D, Gilbody S. Behavioural Activation for Social IsoLation (BASIL+) trial (Behavioural activation to mitigate depression and loneliness among older people with long-term conditions): Protocol for a fully-powered pragmatic randomised controlled trial. PLoS One. 2022 Mar 24;17(3):e0263856. doi: 10.1371/journal.pone.0263856. eCollection 2022. PMID 35324908

DOCUMENTS (1):
  • Study Protocol (2022-12-09): https://cdn.clinicaltrials.gov/large-docs/28/NCT05646628/Prot_001.pdf